CLINICAL TRIAL: NCT06764927
Title: Fibrinogen in Liver Transplant Subjects
Acronym: FITS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ezeldeen Abuelkasem (Other)
Responsible Party: Sponsor-Investigator, Ezeldeen Abuelkasem, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24070113
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Liver Transplant Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, unblinded, randomized controlled study.
Masking Description: N/A - unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Cryoprecipitate Antihemophilic Factor (AHF) (Active Comparator): AHF is the standard of care plasma product often used in liver transplant cases. The procedures to implementing AHF include requesting the order of this plasma product and then waiting for the product to be thawed for use, which can take approximately 10-15 minutes. Subjects assigned to this group will receive all standard of care procedures, including the use of AHF if required during their scheduled surgery.
  Interventions: Biological: Cryoprecipitate Antihemophilic Factor (AHF)
- Investigational Cryoprecipitate Intercept Fibrinogen Complex (IFC) (Active Comparator): IFC is an approved plasma product that is not typically stored in the OR for liver transplant cases. Subjects assigned to this group will receive standard of care procedures, with the addition of IFC being readily available in their designated OR to eliminate any delay if they are to require the use of a plasma product.
  Interventions: Biological: Cryoprecipitate Intercept Fibrinogen Complex (IFC)

INTERVENTIONS:
Biological: Cryoprecipitate Intercept Fibrinogen Complex (IFC) — INTERCEPT Fibrinogen Complex is a pathogen-reduced cryoprecipitated fibrinogen complex derived from human plasma. It contains fibrinogen, Factor XIII, and von Willebrand factor to achieve stable clot formation and restore hemostasis1. Recently approved by the US Food and Drug Administration, it is used for the treatment of bleeding associated with fibrinogen deficiency.
  Arms: Investigational Cryoprecipitate Intercept Fibrinogen Complex (IFC)
Biological: Cryoprecipitate Antihemophilic Factor (AHF) — Cryoprecipitate Antihemophilic Factor (AHF), also known as cryo, is a frozen blood product prepared from blood plasma. It is used for fibrinogen supplementation, particularly for hypofibrinogenemia fibrinogen, anemia associated with bleeding or congenital deficiency.
  Arms: Standard Cryoprecipitate Antihemophilic Factor (AHF)

SUMMARY:
The study is a prospective, multi-centered, unblinded, randomized controlled pilot study. The primary objective is to compare functional hemostatic capacity of Investigational Cryoprecipitate Intercept Fibrinogen Complex (IFC) to Standard Cryoprecipitate Antihemophilic Factor (AHF) for liver transplant patients with bleeding and hypofibrinogenemia to determine impact of earlier access to a concentrated source of fibrinogen in a goal-directed manner.

DETAILED DESCRIPTION:
Fibrinogen is an important factor for hemostasis and when it is deficient or dysfunctional replacing it will improve hemostasis and reduce bleeding. Observational data indicates the use of cryoprecipitate as a source of fibrinogen may reduce bleeding and improve outcomes in patients with severe bleeding. Liver transplant patients often become hypofibrinogenemic and may benefit from early goal directed use of cryoprecipitate or IFC. IFC can be more readily available since it can be stored at room temperature compared to cryoprecipitate which requires thawing. As a result, IFC can be immediately available when indicated compared to the delay in administration of cryoprecipitate due to the need for it to be thawed. This trial will compare clinical outcomes for subjects randomized to either cryoprecipitate or IFC in bleeding liver transplant patients with reduced fibrinogen function.

There is no data comparing outcomes for subjects receiving IFC or cryoprecipitate in any patient population.

The rationale for this trial is to compare IFC to cryoprecipitate (cryo) to assist with the design of a future definitice multicenter trial. Potential advantages of IFC are that since it is stored at room temperature it can be made immediatwlt available whereas with cryo the delay in treatment can be 30 to 40 min due to the need to thaw it from a frozen state. The reduced time to treatment of bleeding may improve outcomes with the use of IFC compared to cryo. In vitro data indicates similar hemostatic function between IFC and Cryo. IFC is pathogen reduced cryoprecipitate. The pathogen reduction methods are licensed for IFC and there has been no safety concerns regarding its use at the centers that are currently using it as their standard product (unpublished).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled to undergo cadaveric liver transplant
* Meets at least one of the following criteria:
* Baseline fibrinogen <200 mg/dL
* Alcoholic cirrhosis
* Nonalcoholic Steatohepatitis (NASH)
* HCV infection

Exclusion Criteria:

* Living related donor transplant
* DCD liver recipient
* Known prothrombotic disorder
* Patient objection to blood transfusion
* Known severe allergic reaction to plasma-based products
* IgA deficiency with known hypersensitivity reaction to plasma
* Hepatocellular/cholangio carcinoma
* Primary biliary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Amount of blood products (24-hours) | 24-hours after initial blood product administration
  The amount of blood products (mL) administered will be collected at the 24-hour timepoint per intervention group and reported as the mean (mL).

SECONDARY OUTCOMES:
Change in TEG parameters | 14 days post-surgery
  Change in TEG parameters, in particular the % change in the alpha angle will be calculated for each study participant and the effect size of the differences in the change, and 95% confidence interval.
Costs of blood products | 14 days post-surgery
  The costs (USD) of blood products used per intervention group will be collected 14-days post-surgery and reported as the mean (USD).
Costs of IV hemostatic agents | 14 days post-surgery
  The costs (USD) of IV hemostatic agents used per intervention group will be collected 14-days post-surgery and reported as the mean (USD).

CONTACTS AND LOCATIONS:
Overall Officials: Ezeldeen Abuelkasem, MBBCh, MSc, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Cincinnati, Cincinnati, Ohio
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data from the participating site, University of Cincinnati College of Medicine, will be shared with Pitt.
  In the future, the investigators may decide to share data with other investigators both within and outside of the institution. If this were to occur, we would de-identify all of the information prior to sharing data in this way. The Office of Sponsored Programs will be contacted prior to sharing data to determine if a date use agreement is necessary.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD sharing will occur up to the anticipated study completion in March 2026
Access Criteria: IRB-approved investigators at the University of Pittsburgh will be the only research personnel with access to all of the IPD and supporting information.